CLINICAL TRIAL: NCT01097148
Title: Peri -and Postoperative Drug Therapy Schedules for Morbidly Obese Patients
Acronym: POP-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: S. van Kralingen, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: V.09.231/R-09
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2009-11

CONDITIONS: Obese; Atracurium; Cefazolin; Morphine; Nadroparin
Keywords: Obese; Atracurium; Cefazolin; Morfine; Nadroparin
MeSH Terms: conditions — Obesity | interventions — Atracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Atracurium, TBW (Active Comparator): Dose of atracurium 0.5 mg/kg based on total body weight
  Interventions: Drug: Atracurium, TBW
- Atracurium IBW (Active Comparator): dose 0.5 mg/kg based on ideal body weight
  Interventions: Drug: Atracurium, TBW

INTERVENTIONS:
Drug: Atracurium, TBW — Dose atracurium 0.5 mg/kg based on total body weight

SUMMARY:
Rationale: Obesity is an increasing health risk worldwide, with the USA recording prevalence in adults of around 20%. The mean body weight of obese patients is also increasing. One of the strategies to treat extreme obesity (Body Mass Index (BMI) > 40 kg/m2) is weight-reducing surgery like laparoscopic gastric banding or gastric bypass. During anaesthesia, morbidly obese patients are exposed to an increased risk at developing postoperative wound infections, apnoea and thrombotic events and may be more difficult to intubate. Routinely, amongst others, cefazolin, morphine, nadroparin and atracurium are administered in standard dosages. However, it is not known to what extend the pharmacokinetics and/or -dynamics of these drugs are affected in morbidly obese patients. Therefore, evidence-based dosing schedules for these drugs in morbidly obese patients should be developed.

Objective: The study is performed in order to develop population pharmacokinetic and/or pharmacodynamic models of the routinely used drug therapies during bariatric surgery in morbidly obese patients (BMI > 40 kg/m2): cefazolin, morphine, nadroparin and atracurium.

A covariate analysis will be performed in order to account for variability in pharmacokinetic and/or pharmacodynamic parameters. This covariate analysis will take into account procedure and patient bound covariates, with specific interest for body weight as a covariate. Whenever possible, non-obese patients will be included in the covariate analysis.

The results will be used to develop individualised dosing schemes for routinely used drugs peri-operatively in morbidly obese patients.

Study design: A randomised, prospective, observational, therapeutic and invasive study.

Study population: Morbidly obese patients with a Body Mass Index > 40 kg/m2 undergoing laparoscopic banding or gastric bypass surgery, 18-60 years old. A total of 20 patients will be included in the study.

Intervention (if applicable): All measurements and data collection will take place around administration of drugs that are given according to routine clinical practice (cefazolin 2 grams for prophylaxis of infections, morphine 10 mg intravenously at the end of surgery, a patient-controlled analgesia (PCA) pump with morphine for postoperative pain relief and nadroparin 0,6 ml for trombo-embolic prophylaxis). For muscle relaxation, patients are randomised to receive one of two generally accepted dosing regimen of atracurium (0.5 mg/kg based on ideal body weight or 0.5 mg/kg based on total body weight). Peri- and postoperatively, a maximum amount of 70 ml of blood will be collected from an indwelling arterial line for measurement of concentrations of cefazolin, morphine, and anti-Xa (nadroparin). One week after surgery the patient will be checked for thrombosis using ultrasonography.

Main study parameters/endpoints:

Primary endpoints to evaluate in morbidly obese patients are;

* pharmacokinetic parameters of cefazolin in blood;
* pharmacokinetic parameters of morphine and metabolites in blood;
* time course of anti-factor Xa levels in blood following nadroparin;
* time course of the pharmacodynamic effect of atracurium.

Secondary endpoints to evaluate in morbidly obese patients are:

* to compare primary endpoints (obtained in morbidly obese patients) with data of non-obese patients
* the occurrence of postoperative wound infections;
* postoperative pain scores, sedation scores and nausea scores;
* the occurrence of bleedings or thrombotic events ;
* required amounts of morphine (PCA);
* to compare the time course of the pharmacodynamic effect of two different doses of atracurium.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients undergoing bariatric surgery with a BMI > 40 kg/m2, ASA I-III

Exclusion Criteria:

* Epilepsy, pregnancy, breastfeeding and known allergy allergies to cefazolin, morphine, nadroparin, atracurium, or benzene sulphonic acid. History of coagulation disorder or history of heparin/LMWH induced thrombocytopenia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Time course of the pharmacodynamic effect of atracurium | 6 months
Pharmacokinetic parameters of cefazolin in blood | 6 months
Pharmacokinetic parameters of morphine and metabolites in blood | 6 months
Time course of anti-factor Xa levels in blood following nadroparin | 6 months

SECONDARY OUTCOMES:
Dosing of atracurium based on total or ideal body weight | 6 months
To compare primary endpoints (obtained in morbidly obese patients) with data of non-obese patients | 6 months
The occurrence of postoperative wound infections | 6 months
Postoperative pain scores, sedation scores and nausea scores | 6 months
The occurrence of bleedings or thrombotic events | 6 months
Required amounts of morphine (PCA) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Simone van Kralingen, MD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Netherlands

REFERENCES:
- [Derived] de Hoogd S, Valitalo PAJ, Dahan A, van Kralingen S, Coughtrie MMW, van Dongen EPA, van Ramshorst B, Knibbe CAJ. Influence of Morbid Obesity on the Pharmacokinetics of Morphine, Morphine-3-Glucuronide, and Morphine-6-Glucuronide. Clin Pharmacokinet. 2017 Dec;56(12):1577-1587. doi: 10.1007/s40262-017-0544-2. PMID 28510797
- [Derived] Diepstraten J, Janssen EJ, Hackeng CM, van Dongen EP, Wiezer RJ, van Ramshorst B, Knibbe CA. Population pharmacodynamic model for low molecular weight heparin nadroparin in morbidly obese and non-obese patients using anti-Xa levels as endpoint. Eur J Clin Pharmacol. 2015 Jan;71(1):25-34. doi: 10.1007/s00228-014-1760-4. Epub 2014 Oct 12. PMID 25304008